CLINICAL TRIAL: NCT05533242
Title: A Phase I Trial to Determine the Maximum Tolerated Dose and Patient-specific Dosimetry of Fractionated Intracavitary Radioimmunotherapy with Lu-177 Labeled 6A10 Fab-fragments in Patients with Glioblastoma After Standard Treatment
Brief Title: Radioimmunotherapy with Lu-177 Labeled 6A10 Fab-fragments in Patients with Glioblastoma After Standard Treatment
Acronym: RIT in GBM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Isotope Technologies Munich (ITM) Oncologics (Unknown); Helmholtz Zentrum München Deutsches Forschungszentrum für Gesundheit und Umwelt (GmbH) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UKM15_0027
Record Dates: First submitted 2022-07-25; First posted 2022-09-08 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Glioblastom WHO Grade 4
Keywords: Carbonic anhydrase XII (CA XII); Intracavitary radioimmunotherapy; Fab fragment 6A10

STUDY DESIGN:
Intervention Model Description: A modified 3+3 design is used. The applied dose of Lu-177-labeled-6A10Fab-fragments to the resection cavity will be escalated in three cohorts until the maximum tolerated dose (MTD) is determined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lu-177-labeled-6A10Fab-fragments (Experimental): The patient will receive a predetermined dose of Lu-177-labeled- 6A10Fab-fragments via the intracavitary reservoir. Patients will receive 3 RIT-cycles with an interval of 4 weeks. The total activity, adjusted to the volume of the RC, will be injected in 3 fractions with 50%, 25% and 25% of the total activity to achieve the desired boost to the 2 cm margin.
  Interventions: Drug: Lu-177 labeled 6A10-Fab-fragments

INTERVENTIONS:
Drug: Lu-177 labeled 6A10-Fab-fragments — The antibody 6A10 is a specific CA12 Inhibitor, a highly specific glioma cell-associated enzyme; all tumor cells are CA12-positive, while its expression in normal brain is very low, and Lu-177 has a comparable β-emission, but a significantly low γ-Emission.

SUMMARY:
Locoregional, intracavitary radioimmunotherapy (iRIT) with a newly developed radioimmunoconjugate (Lu-177 labeled 6A10-Fab-fragments) will be used to prevent or postpone tumour recurrence in patients with GBM following standard therapy .

Following study objectives will be analyzed:

* Determining the Maximum Tolerated Dose (MTD)
* Determining safety by assessing all new neurological, hematological and other AEs CTC grade 2 or higher
* Determining absorbed dose to the 2 cm shell of the resection cavity (based on a series of SPECT/CTs of the head 2h,24h,48h, 72h p.i. and on day 5-7)
* Determining absorbed dose values for the kidneys, the liver, the active marrow (based on a series of SPECT/CTs of the abdomen 2h,24h,48h, 72h p.i. and on day 5-7)
* Determining 24 weeks Progression-Free-Survival (PFS), defined from the day of inclusion

DETAILED DESCRIPTION:
In glioblastoma (GBM), tumour recurrence occurs adjacent to the initial tumor resection cavity in about 85% of cases (Albert et al., 1994; Bashir et al., 1988; Nestler et al., 2015). Therefore, local treatment concepts seem crucial for effective recurrence treatment strategies. We consider locoregional, intracavitary radioimmunotherapy (iRIT) to be a new therapeutic approach to delay or prevent the development of local tumour regrowth in GBM patients. By applying a radioimmunoconjugate (RIC) into the surgically created resection cavity (RC) the blood-brain barrier can effectively be by-passed, allowing the a deposit of high radiation doses locally while sparing sensitive organs like the bone marrow and the kidneys. LuCaFab (Lu-177 labeled 6A10- Fab-fragment) is a carbonic anhydrase XII-specific antibody Fab fragment developed by Helmholtz Munich, labeled with ITM's highly pure medical radioisotope, lutetium-177. (ITM IsotopeTechnologies Munich SE). Patients with GBM after standard therapy (surgery by radio-chemotherapy concomitant and adjuvant chemotherapy) Are eligible for the study. Patients will receive the calculated total doses of Lu-177-labeled 6A10-Fabs in three fractions with an interval of 4 weeks between injections, administered into the tumour cavity via an implanted reservoir. A patient specific dosing strategy will be applied and will depend on the individual RC volume. This investigator-initiated trial is sponsored by the University Hospital Münster, conducted in hospitals in Münster, Essen, Cologne, and Wuerzburg, and supported by ITM and Helmholtz Munich.

ELIGIBILITY:
Inclusion Criteria:

* Written patient consent after comprehensive information
* Age between 18 and 80 years
* Primary supratentorial high grade glioma after standard therapy (fluorescence-guided surgery, radio-chemotherapy, concomitant + adjuvant chemotherapy), with no or stable small tumor residue (residual contrast enhancement of up to 5cm3) at earliest 6 weeks after completion of radiotherapy
* Histological verification of glioblastoma and CA 12-expression of tumor cells confirmed
* Karnofsky-score ≥ 60
* Volume of resection cavity 2,5-25 cm3
* Male and female patients with reproductive potential must use an approved contraceptive method
* Pre-menopausal female patients with childbearing potential: a negative serum pregnancy test must be obtained prior to treatment start
* Adequate bone marrow reserve: white blood cell (WBC) count ≥3000/μl, granulocyte count >1500/μl, platelets ≥100000/μl, hemoglobin ≥ 10 g/dl
* Adequate liver function: bilirubin < 1.5 times above upper limit of normal range (ULN), alanine transaminase (ALT/SGPT) and aspartate transaminase (AST/SGOT) < 3 times ULN. In the case of documented or suspected Gilbert's disease bilirubin < 3 times ULN.
* Blood clotting: INR (=PT) and PTT within acceptable limits according to the investigator
* Adequate renal function: creatinine < 3 times above ULN; eGFR > (or equal) 60 ml/min

Exclusion Criteria:

* Patient unable to undergo imaging by CT, PET or contrast-enhanced MRI for whatever reason (i.e., pacemaker)
* Resection cavity with intraventricular access
* Significant leakage of radioactivity into CSF spaces or ventricles
* Other actively treated invasive malignancy
* Breastfeeding women
* Past medical history of diseases with poor prognosis, e.g., severe coronary heart disease, heart failure (NYHA III/IV), severe and poorly controlled diabetes, immune deficiency, residual deficits after stroke, severe mental retardation, pre-existing neurological diseases except those related to glioblastoma or other serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Any active infection (at the discretion of the investigator)
* Previous participation in a registered clinical trial with therapeutic intervention less than 6 weeks prior to enrolment (date of informed consent)
* Allergy against known constituents of study medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Through study completion, ca 1 ½ years
  Determine maximum tolerated dose (MTD) and safety of adjuvant radio-immunotherapy (RIT) with Lu-177 labeled 6A10-Fab-fragments
Safety of the adjuvant radio-immunotherapy | Through study completion, ca 1 ½ years
  Determining safety by assessing all new neurological, hematological and other AEs CTC grade 2 or higher

SECONDARY OUTCOMES:
Evaluation of pharmacokinetics of Lu-177 labeled 6A10 Fab fragments | After first application: 2 ,24 ,48, 72 hours post injection and on day 5-7. After second and third application.
  Determining absorbed dose to the 2 cm shell of the resection cavity (based on a series of SPECT/CTs of the head 2 ,24 ,48, 72 hours post injection and on day 5-7). Determining absorbed dose values for the kidneys, the liver, the active marrow (based on a series of SPECT/CTs of the abdomen 2 ,24 ,48, 72 hours post injection and on day 5-7)
Progression-free survival (PFS) | Through study completion, an average of 18 months
  Determining 24 weeks Progression-Free-Survival (PFS), defined from the day of inclusion

OTHER OUTCOMES:
Overall survival (OS) | 2 years from the day of inclusion
  OS is defined as the period of time from the start of a study or the treatment in a study until the death of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stummer, Prof., Principal Investigator — University Hospital Muenster, Klinik und Poliklinik für Neurochirurgie
Locations (7):
- Germany (7):
  - Klinik für Allgemeine Neurochirurgie des Universitätsklinikums Köln, Cologne
  - Klinik für Nuklearmedizin des Universitätsklinikums Köln, Cologne
  - Klinik für Neurochirurgie des Universitätsklinikums Essen, Essen
  - Klinik für Nuklearmedizin, Strahlenklinik des Universitätsklinikums Essen, Essen
  - Klinik für Nuklearmedizin der Universität Münster, Münster
  - Universitätsklinikum Würzburg - Neurochirurgie, Würzburg
  - Universitätsklinikum Würzburg - Nuklearmedizin, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiedler L, Kellner M, Gosewisch A, Oos R, Boning G, Lindner S, Albert N, Bartenstein P, Reulen HJ, Zeidler R, Gildehaus FJ. Evaluation of 177Lu[Lu]-CHX-A''-DTPA-6A10 Fab as a radioimmunotherapy agent targeting carbonic anhydrase XII. Nucl Med Biol. 2018 May;60:55-62. doi: 10.1016/j.nucmedbio.2018.02.004. Epub 2018 Mar 4. PMID 29571067
- [Background] Alterio V, Kellner M, Esposito D, Liesche-Starnecker F, Bua S, Supuran CT, Monti SM, Zeidler R, De Simone G. Biochemical and Structural Insights into Carbonic Anhydrase XII/Fab6A10 Complex. J Mol Biol. 2019 Dec 6;431(24):4910-4921. doi: 10.1016/j.jmb.2019.10.022. Epub 2019 Nov 1. PMID 31682835
- [Background] Battke C, Kremmer E, Mysliwietz J, Gondi G, Dumitru C, Brandau S, Lang S, Vullo D, Supuran C, Zeidler R. Generation and characterization of the first inhibitory antibody targeting tumour-associated carbonic anhydrase XII. Cancer Immunol Immunother. 2011 May;60(5):649-58. doi: 10.1007/s00262-011-0980-z. Epub 2011 Feb 5. PMID 21298264
- [Background] Gondi G, Mysliwietz J, Hulikova A, Jen JP, Swietach P, Kremmer E, Zeidler R. Antitumor efficacy of a monoclonal antibody that inhibits the activity of cancer-associated carbonic anhydrase XII. Cancer Res. 2013 Nov 1;73(21):6494-503. doi: 10.1158/0008-5472.CAN-13-1110. Epub 2013 Sep 12. PMID 24030978
- [Background] Proescholdt MA, Mayer C, Kubitza M, Schubert T, Liao SY, Stanbridge EJ, Ivanov S, Oldfield EH, Brawanski A, Merrill MJ. Expression of hypoxia-inducible carbonic anhydrases in brain tumors. Neuro Oncol. 2005 Oct;7(4):465-75. doi: 10.1215/S1152851705000025. PMID 16212811
- [Background] Supuran CT. Carbonic anhydrase inhibitors as emerging agents for the treatment and imaging of hypoxic tumors. Expert Opin Investig Drugs. 2018 Dec;27(12):963-970. doi: 10.1080/13543784.2018.1548608. Epub 2018 Nov 22. PMID 30426805